CLINICAL TRIAL: NCT07103616
Title: Individual Cerebral Hemodynamic Oxygenation Relationships - ICHOR 4
Acronym: ICHOR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Matthew Borzage, Assistant Professor of Research Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CHLA-25-00084; 5K25HL153954-03 (NIH)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia; Reaction; Anesthesia
Keywords: Magnetic Resonance Imaging; Cerebral Blood Flow; Cerebral Metabolism; Anesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participant and care provider will be aware randomization status. Investigator and outcomes assessor will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Propofol (Experimental): Subject will receive propofol anesthesia during their MRI. Dosage form: injectable solution. Dosage: 100-300 mcg/kg/min, or as per clinical standard of care appropriate for specific subjects.
  Frequency and duration: continuous infusion while undergoing MRI.
  Interventions: Drug: Randomization of Propofol or Dexmedetomidine
- Dexmedetomidine (Experimental): Subject will receive Dexmedetomidine during their MRI. Dosage form: injectable solution. Dosage: Generally, initiate at 0.6 mcg/kg/hour and titrate to achieve desired clinical effect with dosages ranging from 0.2 to 1 mcg/kg/hour or as per clinical standard of care appropriate for specific subjects.
  Frequency and duration: continuous infusion while undergoing MRI.
  Interventions: Drug: Randomization of Propofol or Dexmedetomidine

INTERVENTIONS:
Drug: Randomization of Propofol or Dexmedetomidine — This intervention is a randomization of Propofol or Dexmedetomidine. Each group will receive three minutes of research images, followed by induction of anesthesia and immediately followed by three minutes of imaging. The subject will receive standard care clinical magnetic resonance imaging for 45 minutes and three minutes of research images at the end of the scan.

SUMMARY:
The goal of this clinical trial is to understand whether there are differences in the cerebral blood flow, and oxygen metabolism affected by two types of anesthesia: Propofol or Dexmedetomidine. Subjects who require clinical anesthesia for a clinical MRI and for whom the use of Propofol and Dexmedetomidine are in clinical equipoise will be offered to have the anesthesia they will receive during their MRI randomized.

* Change in cerebral blood flow (ml blood/100g/min)
* Change in cerebral metabolic rate of oxygen (ml O2/100g/min)

Researchers will compare Propofol (Group A) to Dexmedetomidine (Group B) to see if compare the hemodynamic response to anesthesia.

Participants will be randomized to receive one of two equally safe anesthetics (Propofol or Dexmedetomidine).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for a clinically indicated MRI at the sponsor institution.
* Patients who are able to tolerate an MRI.
* Patients who require clinical anesthesia for their MRI.
* Patients with conditions not believed to alter oxygen metabolism or blood flow in the brain, including but not limited to patients with orthopedic indications, undescended testicles, hernia repairs, term equivalent age scans.
* Patients who have no medical conditions that make the use of propofol or dexmedetomidine better for their clinical outcome.
* Patients between birth and up-to 7 year of age.
* Patients with conditions known to alter oxygen metabolism or blood flow in the brain, e.g. traumatic brain injury, hypoxic ischemic encephalopathy, tumor.

Exclusion Criteria:

* Patients with an MRI-incompatible device or implant (e.g. pacemakers, stents)
* Preterm infants less than 25 weeks postmenstrual age (PMA) at the time of the scan.
* Patients who are clinically too unstable to extend their MRI by up-to 10 minutes.
* Patients who do not require clinical anesthesia.
* Patients at risk for propofol infusion syndrome (known severe metabolic acidosis, hyperkalemia, lipemia, rhabdomyolysis, hepatomegaly, renal failure, ECG ST segment elevation, and/or cardiac failure)
* Patient at risk for sensitivity to volatile halogenated anesthetic agents (known congenital Long QT Syndrome or patients taking drugs that can prolong the QT interval),
* Patients with Perioperative Hyperkalemia (known neuromuscular disease, particularly Duchenne muscular dystrophy)

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral blood flow (ml blood/100g/min) | Time points over which the change is assessed: change from (1) start of MRI, (2) after induction of anesthesia, (3) MRI completion, an average of 60 minutes.
  Phase contrast (PC) acquisition via MRI will be used to assess any impact of anesthesia on cerebral blood flow.
Change in cerebral metabolic rate of oxygen (ml O2/100g/min) | Time points over which the change is assessed: change from (1) start of MRI, (2) after induction of anesthesia, (3) MRI completion, an average of 60 minutes
  T2 relaxation under spin tagging (TRUST) acquisition via MRI will be used to assess any impact of anesthesia on cerebral metabolic rate of oxygen.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Borzage, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No